CLINICAL TRIAL: NCT04651881
Title: A Randomized, Open-label, Single Dose, Crossover Study to Investigate the Pharmacokinetic Profiles and Safety of High-dose CKD-385 in Healthy Volunteers Under Fed Conditions
Brief Title: Clinical Study to Investigate the PK Profiles and Safety of CKD-385 in Healthy Volunteers Under Fed Conditions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A88_09BE2016P
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Experimental): 1. Period 1: Reference drug
  2. Period 2: Test drug 1
  3. Period 3: Test drug 2
  Interventions: Drug: Reference drug; Drug: Test drug 1; Drug: Test drug 2
- Group 2 (Experimental): 1. Period 1: Test drug 2
  2. Period 2: Reference drug
  3. Period 3: Test drug 1
  Interventions: Drug: Reference drug; Drug: Test drug 1; Drug: Test drug 2
- Group 3 (Experimental): 1. Period 1: Test drug 1
  2. Period 2: Test drug 2
  3. Period 3: Reference drug
  Interventions: Drug: Reference drug; Drug: Test drug 1; Drug: Test drug 2
- Group 4 (Experimental): 1. Period 1: Test drug 2
  2. Period 2: Test drug 1
  3. Period 3: Reference drug
  Interventions: Drug: Reference drug; Drug: Test drug 1; Drug: Test drug 2
- Group 5 (Experimental): 1. Period 1: Test drug 1
  2. Period 2: Reference drug
  3. Period 3: Test drug 2
  Interventions: Drug: Reference drug; Drug: Test drug 1; Drug: Test drug 2
- Group 6 (Experimental): 1. Period 1: Reference drug
  2. Period 2: Test drug 2
  3. Period 3: Test drug 1
  Interventions: Drug: Reference drug; Drug: Test drug 1; Drug: Test drug 2

INTERVENTIONS:
Drug: Reference drug — 1 Cap., single oral administration under fed condition
  Other Names: D744
Drug: Test drug 1 — 1 Tab., single oral administration under fed condition
  Other Names: CKD-385 64 mg formulation I (878mg)
Drug: Test drug 2 — 1 Tab., single oral administration under fed condition
  Other Names: CKD-385 64 mg formulation II (878mg)

SUMMARY:
Clinical Study to Investigate the Pharmacokinetic Profiles and Safety of High-dose CKD-385 in Healthy Volunteers under fed conditions

DETAILED DESCRIPTION:
A randomized, open-label, single dose, crossover study to investigate the pharmacokinetic profiles and safety of high-dose CKD-385 in healthy volunteers under fed conditions

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult aged more than 19 at the time of screening
2. Those who had 18.0kg/m² ≤ Body Mass Index (BMI) < 30.0kg/m²

   # BMI=Weight(kg) / Height(m)²
3. Those who have no congenital diseases or chronic diseases and have no abnormal symptoms or findings on a medical examination.
4. Those who are eligible for clinical trials based on laboratory (hematology, blood chemistry, urinalysis, serology), vital signs and ECG results at screening.
5. Those who have voluntarily given written informed consents to participate in the study and to comply with all the instructions, based on full understanding of the nature of the study after listening to detailed explanations.
6. Those who agree to double contraception method from the 1st dministration of the investigational product until 7 days after the last administration of investigational product.

Exclusion Criteria:

1. Those who has medical evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, urinary, cardiovascular, hepatic, psychiatric, neurologic or allergic diseases(except for simple dental history such as tartar, mpacted teeth, wisdom teeth).
2. Those with a medical history of gastrointestinal disorders(esophageal achalasia or esophagus stenosis, Crohn's disease) or gastrointestinal surgery(except for simple appendicitis surgery or hernia surgery or tooth extraction surgery) that may affect the absorption of drug.
3. Those who has a history of regular alcohol consumption in excess of 14 glasses/week for woman, 21 glasses/week for man within 1 months prior to screening.
4. Those who received investigational products or bioequivalence test drugs within 6 months before the first administration of clinical trial drugs.
5. Those who take drugs which may cause induction or inhibition of drug metabolism within 30 days before the first administration of investigational products.
6. Those who have taken any drugs that may affect the clinical trial within 10 days.
7. Those who donated whole blood within 2 months, or blood components within 2 week before first administration of investigational products.
8. Those who is unable to consume a high-fat meal provided during the study.
9. Those who are deemed insufficient to participate in this clinical study by investigators.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2020-12-09 (Estimated); Study Completion 2020-12-09 (Estimated)

PRIMARY OUTCOMES:
AUCt of CKD-385 | Pre-dose (0 h),1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 8, 10, 12, 24, 48 hours
  Area under the concentration-time curve from time zero to time of CKD-385
Cmax of CKD-385 | Pre-dose (0 h),1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 8, 10, 12, 24, 48 hours
  Maximum plasma concentration of CKD-385

SECONDARY OUTCOMES:
AUCinf of CKD-385 | Pre-dose (0 h),1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 8, 10, 12, 24, 48 hours
  Area under the concentration-time curve from zero up to infinity of CKD-385
Tmax of CKD-385 | Pre-dose (0 h),1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 8, 10, 12, 24, 48 hours
  Time to maximum plasma concentration of CKD-385
T1/2 of CKD-385 | Pre-dose (0 h),1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 8, 10, 12, 24, 48 hours
  Terminal elimination half-life of CKD-385
CL/F of CKD-385 | Pre-dose (0 h),1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 8, 10, 12, 24, 48 hours
  Apparent clearance of CKD-385
Vd/F of CKD-385 | Pre-dose (0 h),1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 8, 10, 12, 24, 48 hours
  Apparent Volume of Distribution of CKD-385

CONTACTS AND LOCATIONS:
Overall Officials: Min-gi Kim, Principal Investigator — CENTRAL HOSPITAL
Locations (1):
- Central Hospital, Gyeonggi-do, Siheung-si, South Korea